CLINICAL TRIAL: NCT05485454
Title: A Pilot Cross-Over Preference Study of Two Pneumatic Compression Devices for Patients With Lower Limb Lymphedema
Brief Title: A Preference Study of Two Pneumatic Compression Devices for Patients With Lower Limb Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Collaborators: Lymphatic Solutions, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AF22-04-01
Record Dates: First submitted 2022-07-18; First posted 2022-08-03 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Lymphedema of Leg; Lymphedema; Lymphedema, Secondary; Lymphedema Primary; Lymphedema, Lower Limb
Keywords: Pneumatic Compression Device
MeSH Terms: conditions — Lymphedema; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Aria Health Aria Free (Active Comparator): An Aria Free therapy session on the study lower limb.
  Interventions: Device: Aria Health Aria Free
- Traditional PCD (Active Comparator): A therapy session using the traditional PCD on the study lower limb.
  Interventions: Device: A Traditional PCD

INTERVENTIONS:
Device: Aria Health Aria Free — An in-clinic therapy session with the Aria Free for a duration of 30 minutes under the direct supervision of the Principal Investigator.
  Arms: Aria Health Aria Free
Device: A Traditional PCD — An in-clinic therapy session with the traditional PCD for a duration of 30 minutes under the direct supervision of the Principal Investigator.
  Arms: Traditional PCD

SUMMARY:
This study will aim to undertake a preference evaluation comparing the Aria Health Aria Free™ to a competitor's device by assessing overall satisfaction and preference of the devices individually and in comparison to one another. Twenty (20) subjects will be enrolled on this study at one study site in Houston, Texas.

DETAILED DESCRIPTION:
This research study is studying the preference of the compact Aria Health Aria Free™ Pneumatic Compression System ('Aria Free,' 'Aria') as a treatment for Lower Limb Lymphedema when compared to a traditional pneumatic compression device. A pneumatic compression device is also known as a 'PCD.' Both PCDs used in this study have been approved by United States Food and Drug Administration (FDA) for the treatment of lower limb lymphedema and are Code E0651 pneumatic compression devices, as defined by the Centers for Medicare & Medicaid Services (CMS) under The Healthcare Common Procedure Coding System (HCPCS) for Durable Medical Equipment (DME). Subjects participating in this study are asked to use each PCD for a short therapy session and then answer a series of questionnaires regarding their experience with the devices.

Participation in this study requires one clinic visit that will last about two (2) hours. At the beginning of the visit, the Investigator will ask each subject a series of questions to collect demographic data, and medical and pneumatic compression device usage history. The Investigator will then ask the subject to 'inspect' (touch and handle) the two PCDs used in this study and ask a few questions about the subject's opinion of the two devices based on this inspection. The Investigator will then guide the subject through completion of two (2) thirty (30) minute therapy sessions, one session using the Aria and the other session using the traditional PCD. The order in which the sessions are completed will be random, like the flip of a coin. Before and after each therapy session, the Investigator will complete a series of measurements and take photographs of the subject's lower limbs. The Investigator will also assess the subject's skin and tissue health after each intervention. Subjects will also be asked to complete questionnaires after each therapy session that will ask about subjective satisfaction with and preference between the two devices. Once the study visit has been completed, the subject will have completed the study and may return to his/her usual standard of care activities for treating his/her lower limb lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients who are ≥ 18 years, mentally able to understand and follow the instructions of the study personnel
* A diagnosis of unilateral or bilateral lower limb lymphedema
* A physician's prescription for use of a pneumatic compression device
* Able to provide written informed consent
* Patient can read and comprehend English
* Study leg must be within fit range of the Aria Free Garment (Ankle Max = 35cm/13.78in; Thigh Max = 80cm/34.49in)

Exclusion Criteria:

* Subject undergoing cancer treatment
* Subject has active lower limb wounds
* Subject is pregnant or trying to become pregnant
* History of pulmonary edema or decompensated congestive heart failure
* Subject has any condition in which increased venous and lymphatic return is undesirable
* Subject has inbuilt electrical stimulator, e.g., cardiac pacemaker
* Acute venous disease (acute thrombophlebitis, acute deep venous thrombosis, acute pulmonary embolism)
* Severe peripheral artery disease (critical limb ischemia including ischemic rest pain, arterial wounds or gangrene)
* Active skin or limb infection/inflammatory disease (acute cellulitis, other uncontrolled skin or untreated inflammatory skin disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-11 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Satisfaction and Preference | Satisfaction and Preference ratings will be assessed during the only study visit: Visit 1/Day 1.
  The primary outcome of this study is to compare levels of subjective ratings of satisfaction and preference measurements after completed sessions with Aria Free and the traditional PCD devices. Each session is 30 minutes in duration. Subjective measures for each device will use an 11-point Likert Scale where a score of 10 is considered very favorable and a score of 0 is very unfavorable.

SECONDARY OUTCOMES:
Limb Volume Measurements | Limb volume measurements will be collected during the only study visit: Visit 1/Day 1.
  The Principal Investigator will collect pre and post intervention circumferential limb measurements for each subject and these measurements will be used in a truncated cone formula to calculate total limb volume. Each intervention is 30 minutes in duration. The pre and post total limb volume measurements will be compared and assessed for change.
Clinician's Skin and Tissue Health Assessment | The skin and tissue will be assessed during the only study visit: Visit 1/Day 1.
  The Principal Investigator will assess the skin and tissue health of the study lower limb after each intervention. Each intervention is 30 minutes in duration. Twenty observations are listed for the Investigator to document 'Yes' or 'No' if any of the observations are present or not, respectively, during the lower limb physical exam.

CONTACTS AND LOCATIONS:
Overall Officials: Denise M Baylor, CLT-LANA, Principal Investigator — Lymphatic Solutions, Owner
Locations (1):
- Lymphatic Solutions, LLC, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data available will not be shared with other researchers.